CLINICAL TRIAL: NCT01915355
Title: Pulsed Dye Laser Treatment of Onychomycosis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Thomas Jefferson University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB 13D.230
Record Dates: First submitted 2013-07-29; First posted 2013-08-02 (Estimated); Last update posted 2016-08-19 (Estimated); Status verified 2016-08

CONDITIONS: Onychomycosis
Keywords: onychomycosis; nail; fungus
MeSH Terms: conditions — Onychomycosis | interventions — Lasers, Dye

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Pulsed Dye Laser for fungus treatment (Experimental): The purpose of this research is to investigate the use of the Candela V-beam Pulsed Dye Laser for the treatment of onychomycosis, a common nail fungus.
  Interventions: Device: Pulsed Dye Laser for the treatment of nail fungus

INTERVENTIONS:
Device: Pulsed Dye Laser for the treatment of nail fungus — The purpose of this research is to investigate the use of the Candela V-beam Pulsed Dye Laser for the treatment of onychomycosis, a common nail fungus.

SUMMARY:
The purpose of this research is to investigate the use of the Candela V-beam Pulsed Dye Laser for the treatment of onychomycosis, or nail fungus.

Hypothesis: Complete nail clearance will occur in approximately half of patients after 3 laser treatments.

DETAILED DESCRIPTION:
10 patients will participate nationally. The investigators hope to enroll all 10 patients at Jefferson. Involvement in the study will last about 8-12 weeks for the subject. The entire study will take about 12 months to complete.

ELIGIBILITY:
Inclusion Criteria:

* Ages 18-65 years old
* Diagnosis of onychomycosis based on positive fungal culture for dermatophyte and positive PAS from toenail clipping

Exclusion Criteria:

* HIV/immunosuppression
* Candidal toenail infection
* Prior PO antifungal therapy within last 6 months
* Personal history of psoriasis, lichen planus, or significant photosensitivity disorder
* Any serious generalized medical condition

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2013-07; Primary Completion 2014-12 (Actual); Study Completion 2015-07 (Actual)

PRIMARY OUTCOMES:
Total Nail Clearance | approximately 12 weeks
  After 3 laser treatments, the subject should experience clinical clearance.

CONTACTS AND LOCATIONS:
Overall Officials: Nazanin Saedi, MD, Principal Investigator — Jefferson Dermatology Associates
Locations (1):
- Jefferson Dermatology Associates, Philadelphia, Pennsylvania, United States